







## **ARC Participant Information and Consent Form-Interview**

<u>Title of Study</u>: ARC – Access to Resources in the Community/ Accès aux ressources communautaires

### Principal Investigator (PI) Simone Dahrouge, PhD 613-562-6262 ext. 2913

## **Funding Agencies**:

Canadian Institutes of Health Research SPOR initiative

Participation in this study is voluntary. Please read this Informed Consent Form carefully before you decide if you will take part. You may also ask the study team as many questions as you like.

#### Why am I being given this form?

You have recently completed a research study about improving access to community resources for patients; the Access to Resources in the Community (ARC) study.

This form asks if you agree to speak with a member of the study team about your experiences while participating in this study. It is up to you if you take part in the interview.

#### Why is this interview being done?

The interview will help the research team know more about your experiences with the services provided to you as a participant in this study. You would be asked about what has helped you or prevented you from going to the community program, and if you went, your experience with using that program.

#### What do I have to do?

The interview would be at a time and place that is easy for you and will take about 45 minutes. It may be done in person or by phone, depending on your preference.

You can refuse to answer any question during the interview.

Whether you choose to participate in the interview or choose not to, it will not change the care you receive from your doctor.

With your permission, the interview will be audio recorded to ensure we have properly captured your answers. If you do not want to be audio recorded, you can still participate in the interview.

#### What are the risks involved in taking part in the interview?

The risks are minimal. You might find the interview is long or that the questions feel personal. You might not like all of the questions that you are asked. You do not have to answer any questions that make you uncomfortable.

#### Can I expect to benefit from participating in this interview?

There is no direct benefit to you in taking part in the interview. By taking part in the interview, you will help the study team better understand whether the navigation services offered in this study help patients make use of programs that can help improve their health and wellbeing.

#### Do I have to take part in the interview?

The decision to take part in the interview is entirely up to you. Whether you choose to take part, or choose not to, it will not change the care you receive from your doctor.







If you choose to participate and change your mind, you may withdraw at any time, and if you wish, all the information that you have provided will be removed and will not use it in the study.

You do not have to answer any question you do not want to.

#### How will my personal information be protected?

The interview file will be identified by a study participant ID only and not by any information that may identify you, such as your name. The link between your participant ID and name will be kept securely and separately from the study data.

If you agree to be audiotaped, the audio recordings will be sent to professional to produce a written document of the interview. Any information that could identify you, such as your name, will be not be included in the study data. Your information will only be identified by your study ID. Only the study team and the professional producing the written document of the interview will have access to the audio recording and written form of the interview.

Study data will be kept by the study team for ten years – this is the same for all studies. After ten years, your information will be safely deleted and destroyed.

#### Who can I call if I have questions?

If you have any questions or should you no longer wish to remain a part of the ARC study, please call Andrea Perna (613) 562-6262 ext.2920 or email <a href="mailto:arc@bruyere.org">arc@bruyere.org</a>. In Sudbury, please call Patrick Timony (705) 675-1151 ext. 4298 or email <a href="mailto:Pe Timony@laurentian.ca">Pe Timony@laurentian.ca</a>

You can also contact the study principal investigator, Simone Dahrouge at (613) 562-6262 ext. 2913 or sdahrouge@bruyere.org. In Sudbury, please contact Alain Gauthier at (705) 675-1151 ext. 4301 or email agauthier@laurentian.ca

The Ottawa Health Science Network Research Ethics Board (OHSN-REB), Bruyère Research Ethics Board, the Hôpital Montfort Research Ethics Board, the University of Ottawa Research Ethics Board, the Laurentian University Research Ethics Board and University of Ontario Institute of Technology have reviewed this protocol. These Boards consider the ethical aspects of all research studies involving human participants at participating hospitals, institutes and universities.

If you have any questions about your rights as a study participant or about the conduct of this study, please contact:

- Chairperson, OHSN-REB at 613-798-5555, ext. 16719
- Research Ethics Coordinator, Bruyère Research Ethics Board at reb@bruyere.org or 613-562-6262 ext. 4003
- Montfort Hospital Research Ethics Board, 745A suite 102 Montreal road, Ottawa, Ontario at 613-746-4621, ext. 2221 or via email at <a href="mailto:ethique@montfort.on.ca">ethique@montfort.on.ca</a>
- Protocol Officer for Ethics in Research, University of Ottawa, <u>at ethics@uottawa.ca</u> or 613-562-5387
- Research Ethics Officer, Laurentian University at 705-675-1151 ext 3213, 2436 or toll free at 1-800-461-4030 or email <a href="mailto:ethics@laurentian.ca">ethics@laurentian.ca</a>.
- Ethics and Compliance Officer, University of Ontario Institute of Technology, researchethics@uoit.ca or 905-721-8668 X 3693







# Access to Resources in the Community - Accès aux ressources communautaires

| ~ | T | | | . • |
|------------|-----------|---------|----------------|----------|
| Consent to | . Vantiai | nata in | an In | tawamaan |
| t omsem n | | пите пп | <b>711 III</b> | iei view |

| <ul> <li>I understand that I am being asked<br/>about my experience with the stud</li> </ul> | d to take part in an interview at the end only | of the ARC study to talk |
|---|---|---|
| •told n | ne about the study. | |
| • I read each page of this form, or h | ad this form read to me. | |
| • All of my questions were answere | ed so that I understand the study. | |
| • I can decide at any time that I do | not want to take part in this interview. | |
| • I have decided to take part in this | interview. | |
| • I will get a copy of this signed for | m. | |
| To indicate consent to the option of b I agree to have my intervie | eing audio recorded <u>please initial in th</u><br>w audio recorded. | e box below: |
| Participant's Printed Name | Participant Signature | Date |
| Verbal consent obtained by | Research Assistant | Date |
| Your Printed Name (Participant) | Participant Signature | Date |
| | to the participant. To the best of my s and benefits involved in taking part in Investigator/Delegate's Signature. | this study. |